CLINICAL TRIAL: NCT03333278
Title: The VitamIn C, HydrocorTisone and ThiAMINe in Patients With Septic Shock Trial (VITAMINS Trial) - A Prospective, Feasibility, Pilot, Multi-centre, Randomised, Open-label Controlled Trial
Brief Title: The Vitamin C, Hydrocortisone and Thiamine in Patients With Septic Shock Trial
Acronym: VITAMINS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Melbourne Health (Other); Barwon Health (Other Government); Monash Health (Other); The Alfred (Other); Wellington Hospital (Other Government); Western Health, Australia (Other Government)
Responsible Party: Principal Investigator, anzicrc, Professor Rinaldo Bellomo, Australian and New Zealand Intensive Care Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC17Austin238
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Shock, Septic; Critically Ill; Vasoplegic Syndrome; Sepsis
Keywords: Critical Care; Shock, Septic; Ascorbic Acid; Adult
MeSH Terms: conditions — Shock, Septic; Critical Illness; Vasoplegia; Sepsis | interventions — Ascorbic Acid; Thiamine; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Multi-centre, Randomised, Open-label controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamins (Active Comparator): intravenous: Ascorbic acid (Vitamin C: 1.5g every 6 hours) Thiamine (Vitamin B1: 200mg every 12 hours) Hydrocortisone (50mg every 6 hours)
  Interventions: Drug: Vitamin C; Drug: Thiamine; Drug: Hydrocortisone,
- Control (Other): Hydrocortisone (50mg every 6 hours)
  Interventions: Drug: Hydrocortisone,

INTERVENTIONS:
Drug: Vitamin C — Ascorbic acid 1.5g every 6 hours i.v. while in ICU, until shock resolution for a maximum of ten days
  Other Names: Ascorbic acid
  Arms: Vitamins
Drug: Thiamine — Thiamine 200mg every 12 hours i.v. while in ICU, until shock resolution for a maximum of ten days
  Other Names: Vitamin B1
  Arms: Vitamins
Drug: Hydrocortisone, — Hydrocortisone 50mg every 6 hours i.v while in ICU, until shock resolution or for a maximum of 7 days, then tapered or stopped.
  Other Names: Solu Cortef

SUMMARY:
Sepsis has been characterised as a dysregulated host response to infection. Adjunctive therapies targeting the inflammatory cascade are being increasingly explored, although to date, have failed to demonstrate consistent benefit, and sepsis continues to manifest poor outcomes. Hospital mortality in patients with septic shock remains as high as 22% in Australia and New Zealand. From a global perspective, 31 million sepsis and 19 million severe sepsis cases are expected to be treated in hospitals all over the world per year.

To date, experimental data have reported that both high dose intravenous vitamin C and corticosteroids attenuate the acceleration of the inflammatory cascade and possibly reduce the endothelial injury characteristic of sepsis, enhance the release of endogenous catecholamines and improve vasopressor responsiveness.

Therefore, the investigators plan to conduct a feasibility pilot prospective, multi-centre, randomised, open-label, trial in ICU patients with septic shock to test whether the intravenous administration of high dose Vitamin C (6g/d), Thiamine (400mg/d) and Hydrocortisone (200mg/d) leads to a more rapid resolution shock and vasopressor dependence.

DETAILED DESCRIPTION:
The investigators plan to conduct a feasibility pilot prospective, multi-centre, randomised, open-label, trial in ICU patients with septic shock to test whether the intravenous administration of high dose Vitamin C (6g/d), Thiamine (400mg/d) and Hydrocortisone (200mg/d) for a maximum of ten days leads to a more rapid resolution shock and vasopressor dependence.

Hypothesis:

Treatment with a combination of intravenous Vitamin C, Thiamine and Hydrocortisone reduces duration of vasopressor (measured by hours alive and vasopressor free) use censored at 7 days compared to standard care with Hydrocortisone alone.

This is a prospective, feasibility, pilot, multi-centre, randomised, open-label controlled trial. This study will be performed in seven Victorian ICUs in Australia. Patients admitted to an ICU of the participating hospitals with the primary diagnosis of septic shock will be screened for inclusion into this study.

Rationale:

Experimental data have demonstrated that both corticosteroids and intravenous vitamin C attenuate the release of pro-inflammatory mediators, reduce the endothelial injury characteristic of sepsis (thereby reducing endothelial permeability and improving microcirculatory flow), augment the release of endogenous catecholamines and enhance vasopressor responsiveness. In animal models, these effects have resulted in reduced organ injury and increased survival. However, their effect in critically ill humans is unknown.

Previous research suggests that vitamin C and glucocorticoids may act synergistically and improve vasopressor responsiveness in patients with sepsis and septic shock.

Randomisation:

ICU patients will be enrolled as soon as possible but no later than 24 hours after fulfilling the criteria for septic shock. Patients will be allocated in a 1:1 ratio to either the treatment group, receiving intravenous Vitamin C (1.5g every 6 hours), Thiamine (200mg every 12 hours) and Hydrocortisone (50mg every 6 hours), or to the control group, receiving Hydrocortisone (50mg every 6 hours) alone.

Treatment allocation will occur using a computerized system and concealed allocation. The clinical staff involved in patient care will administer the additional drugs to those allocated to the treatment arm of the trial as soon as possible after the identification of septic shock and randomization.

Patients readmitted to ICU during the same hospital stay will not receive any further doses of study drugs.

Study Treatment will continue until:

* Septic shock resolves
* The patient leaves the ICU
* Contraindications to Vitamin C, Thiamine or Hydrocortisone therapy arise
* Death occurs
* A maximum of 10 days of treatment has been administered
* Serious adverse events suspected to be secondary to the intervention therapy develop.

Study Drugs

This study will be an open label study:

Intervention group:

* 1500mg Vitamin C is will be diluted in 100ml of Normal Saline (0.9% NaCl) and infused over 1 hour. The dosing schedule is 1500mg every 6 hours for the duration of study treatment.
* 200mg Thiamine will be diluted in 100ml of Normal Saline (0.9% NaCl) and infused over 1 hour. The dosing schedule is 200mg every 12 hours. Patients in the control group of the study can receive thiamine if clinically indicated at the discretion of the attending ICU staff specialist.

In both groups (treatment and control), patients will be treated with hydrocortisone 50mg IV q 6 hourly for the duration of study treatment. After shock resolution and/or a maximum fo 7 days Hydrocortisone will be tapered off or stopped.

Statistical analysis:

Originally, the investigators assumed a mean (SD) duration of vasopressor dependency of 50 (28) hours and estimated a required sample size of 120 patients (60 per group) to identify a clinically relevant decrease of vasopressor dependency and an increase in days alive and vasopressor free at 7 days of 25% (20 hours) (i.e. increase from 41 to 55 hours of days alive and vasopressor free at day 7) with a power of 90% at an alpha level of 0.05.

The investigators have recalculated the sample size based on the pooled standard deviation of hours alive and vasopressor free of the first 59 participants. The pooled standard deviation of hours alive and vasopressor free at 7 days for the 59 patients is 51.6 hours.

To have a 90% power (2 sided p-value of 0.05) to detect a 25-hour difference based on a standard deviation of 51.6, the trial will require 180 patients (90 per group). Allowing for a 20% inflation for non-normality and dropout/withdrawal, the required total sample size is 216 (108 per group). The robustness of the sample size estimate will be further assessed after recruitment of 108 patients (50% of the sample size).

Consent: The major ethical issues associated with this study relate involve the recruitment of participants who are dependent on medical care and in need of immediate intervention for the management of life-threatening haemodynamic instability.

1. Informed consent from participant or substitute/medical treatment decision maker: Where possible, and as authorised by law, which varies between jurisdictions, consent will be obtained from the participant himself or from the participant's legal surrogate if the patient lacks decision-making capacity.
2. Consent to continue: Where it is not possible or practicable for the patient or the legal surrogate to consider the study and give consent immediately, the patient may be enrolled with a waiver of consent (or medical research procedures in an emergency in Victoria) and consent obtained from the participant's legal surrogate as soon as possible, provided the procedure is in accord with the requirements of the site's Human Research Ethics Committee (HREC) and applicable legislation. When appropriate, the participant's legal surrogate, and, in turn, the participant, will be informed of the study and will be able to withdraw consent for ongoing participation at any time.
3. Verbal/Telephone consent: In cases where the participant's legal surrogate cannot attend the hospital to sign the consent form within the time constraints of the study, consent for patient participation in the study may be obtained over the telephone in accordance with local HREC guidelines. The telephone conversation must be documented in the patient's medical record. As soon as the participant's legal surrogate is able to attend the hospital, they will be asked to sign a consent form and note that telephone consent was already provided.

Once subjects are recovered and are able to consider the information sheet, they will be offered the opportunity to withdraw from study follow-up. If a participant dies due to the nature of their critical illness before consent was able to be obtained from the person responsible/medical treatment decision maker, then consent will not be sought and data collected will be used. This is in line with the process followed by other similar intensive care studies conducted previously and approved by the relevant HRECs all where consent to continue has been utilised.

ELIGIBILITY:
Inclusion Criteria:

Patient in the intensive care unit (ICU) with septic shock:

* Blood lactate >2 mmol/L, despite adequate fluid resuscitation AND
* need for continuous vasopressor therapy to keep mean arterial pressure (MAP) >65 mmHg for >2 hours

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. DNR (do not resuscitate)/DNI (do not intubate) orders
4. Death is deemed to be imminent or inevitable during this admission, and either the attending physician, patient or substitute decision-maker is not committed to active treatment
5. Patients with known HIV infection
6. Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency
7. Patients transferred from another ICU or hospital with a diagnosis of a septic shock for > 24 hours
8. Patients with a diagnosis of a septic shock for > 24 hours
9. Patients with known or suspected

   * a. history of oxalate nephropathy or hyperoxaluria
   * b. short bowel syndrome or severe fat-malabsorption
   * c. acute beri-beri disease
   * d. acute Wernicke's encephalopathy
   * e. malaria
   * f. scurvy
   * g. Addison's disease
   * h. Cushing's disease
10. Clinician expects to prescribe systemic glucocorticoids for an indication other than septic shock (not including nebulised or inhaled corticosteroid)
11. Patient is receiving treatment for systemic fungal infection or has documented Strongyloides infection at the time of randomisation
12. Patient with known chronic iron overload due to iron storage and other diseases
13. Patient previously enrolled in this study
14. Clinician expects to prescribe high dose vitamin C for another indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Time alive and free of vasopressors at day 7 (168 hours) after randomization. | 7 days (168 hours)
  This is defined by the patient being alive at discontinuation of all vasopressors for at least 4 hours in the presence of a MAP>65 mmHg for the same 4 hour period as recorded in the ICU charts and censored at 7 days. If a patient dies while on vasopressor therapy, in such a patient, the time alive and vasopressor free time will be 0 - This approach will correct for the competing effect of mortality on duration of vasopressor therapy.

SECONDARY OUTCOMES:
ICU mortality | 90 days after randomization
  Patient died during the ICU admission
Alive and ICU-free days at day 28 calculated as the number of days alive and out of the ICU to day 28 | 28 days after randomization
  Alive and ICU-free days calculated as the number of days alive and out of the ICU to day 28
Hospital mortality | 90 days after randomization
  Patient died during the hospital admission
28-day mortality | 28 days after randomization
  Patient died within 28 days after randomization
90-day mortality | 90 days after randomization
  Patient died within 90 days after randomization
Delta of Sequential Organ Failure Assessment (SOFA) score at 72 hours | 72 hours after randomization
  defined as the initial total SOFA* score minus the day three (72 hours) SOFA score
  *total SOFA = Sequential Organ Failure Assessment = sum of each organ system point score. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. The organ scores are ranging from 0-4, with the best score being 0 and the worst being 4 points. The maximal (and worst) total SOFA score is 24 points.
Hospital length of stay | 90 days after randomization
  Duration the patient stayed in the hospital
28 day cumulative vasopressor free hours | 28 days after randomization
  Cumulative vasopressor free hours from shock resolution to day28 post randomisation
28 day cumulative invasive mechanical ventilation free hours | 28 days after randomization
  Cumulative invasive mechanical ventilation-free hours during the 28 day period post randomisation
RRT duration | 28 days after randomization
  Length of renal replacement therapy dependency during the 28 day period post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, Professor, Principal Investigator — Austin Hospital, Melbourne Australia; Nora Luethi, MD, Principal Investigator — ANZIC-RC; Tomoko Fujii, MD, Principal Investigator — ANZIC-RC
Locations (8):
- Australia (6):
  - Monash Health (Monash Medical Centre and Dandenong Hospital), Clayton, Victoria
  - Geelong University Hospital, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Western Health (Footscray & Sunshine Hospital), Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Cancer Institute of the State of São Paulo, São Paulo, Brazil
- Wellington Hospital, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Policy is available from the website.
URL: https://www.monash.edu/__data/assets/pdf_file/0010/1790875/terms_of_ref.pdf

REFERENCES:
- [Derived] Fujii T, Luethi N, Young PJ, Frei DR, Eastwood GM, French CJ, Deane AM, Shehabi Y, Hajjar LA, Oliveira G, Udy AA, Orford N, Edney SJ, Hunt AL, Judd HL, Bitker L, Cioccari L, Naorungroj T, Yanase F, Bates S, McGain F, Hudson EP, Al-Bassam W, Dwivedi DB, Peppin C, McCracken P, Orosz J, Bailey M, Bellomo R; VITAMINS Trial Investigators. Effect of Vitamin C, Hydrocortisone, and Thiamine vs Hydrocortisone Alone on Time Alive and Free of Vasopressor Support Among Patients With Septic Shock: The VITAMINS Randomized Clinical Trial. JAMA. 2020 Feb 4;323(5):423-431. doi: 10.1001/jama.2019.22176. PMID 31950979
- [Derived] Fujii T, Udy AA, Deane AM, Luethi N, Bailey M, Eastwood GM, Frei D, French C, Orford N, Shehabi Y, Young PJ, Bellomo R; VITAMINS trial investigators. Vitamin C, Hydrocortisone and Thiamine in Patients with Septic Shock (VITAMINS) trial: study protocol and statistical analysis plan. Crit Care Resusc. 2019 Jun;21(2):119-125. PMID 31142242